CLINICAL TRIAL: NCT04743141
Title: Phase 3, Multicenter, Open-label Study to Assess the Long-term Safety and Tolerability of Rimegepant for the Acute Treatment of Migraine (With or Without Aura) in Children and Adolescents ≥ 6 to < 18 Years of Age
Brief Title: Long-term Safety Study of Rimegepant in Pediatric Subjects for the Acute Treatment of Migraine
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BHV3000-312; C4951003 (Other: Alias Study Number); 2024-512744-32-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2021-02-04; First posted 2021-02-08 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Acute Treatment of Migraine
Keywords: Long-term safety, acute treatment, migraine, phonophobia, photophobia, nausea, pediatric, children, adolescent
MeSH Terms: conditions — Migraine Disorders; Hyperacusis; Photophobia; Nausea | interventions — rimegepant sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Active (Experimental): rimegepant 75 mg, 50 mg or 35 mg ODT
  Interventions: Drug: Rimegepant (PF-07899801)

INTERVENTIONS:
Drug: Rimegepant (PF-07899801) — Rimegepant 75 mg, 50 mg or 35 mg ODT

SUMMARY:
The purpose of this study is to test the long-term safety of rimegepant in the acute treatment of migraine in children and adolescents (≥ 6 to < 18 years of age).

ELIGIBILITY:
Inclusion Criteria:

1. History of migraine (with or without aura) for ≥ 6 months before Screening.
2. History of 1 to 8 moderate or severe attacks per month during the 2 months prior to screening.
3. 1 or more migraine days requiring treatment during the Observation Phase.
4. Prophylactic migraine medication is permitted if the dose has been stable for at least 12 weeks prior to the Screening Visit.
5. Ability to distinguish between migraine and other types of headaches.
6. Weight > 15 kg. For EU countries only: Participants 12 to < 18 years of age must have a body weight of >25kg.
7. Adequate venous access for blood sampling.
8. Male and female participants 6 to < 18 years of age (participants must not reach their 18th birthday on or before the Baseline visit).

Exclusion Criteria:

1. History of cluster headache or hemiplegic migraine headache.
2. Confounding and clinically significant pain syndrome.
3. Current uncontrolled and/or untreated psychiatric condition for a minimum of 6 months prior to the Screening Visit (lifetime history of psychosis and/or mania are excluded).
4. History of suicidal behavior or at risk of self-harm/harm to others.
5. History of major psychiatric disorder.
6. Current diagnosis or history of substance abuse
7. Reported current use of or tested positive at Screening for drugs of abuse.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 600 (Estimated)
Dates: Start 2021-04-28 (Actual); Primary Completion 2030-07-31 (Estimated); Study Completion 2030-07-31 (Estimated)

PRIMARY OUTCOMES:
The frequency and severity of on-treatment and treatment-emergent adverse events, serious adverse events, adverse events leading to discontinuation, clinically significant lab abnormalities | 58 weeks
  To evaluate the safety and tolerability of rimegepant in children and adolescents (6 to < 18 years of age).

SECONDARY OUTCOMES:
The frequency and severity of hepatic-related adverse events and frequency of hepatic-related adverse events leading to treatment discontinuation | 58 weeks
  To evaluate the frequency and severity of hepatic-related adverse events and the frequency of hepatic-related treatment discontinuations in children and adolescents (6 to less than 18 years of age) treated with rimegepant.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (124):
- United States (114):
  - Perseverance Research Center, LLC, Scottsdale, Arizona
  - Physicians Research Group, Tempe, Arizona
  - Advanced Research Center, Inc., Anaheim, California
  - ProScience Research Group, Culver City, California
  - Neuro-Pain Medical Center, Fresno, California
  - University of California San Diego, Altman Clinical and Translational Research Institute Clinic, La Jolla, California
  - Adult & Child Neurology Medical Associates, Long Beach, California
  - Memorialcare Miller Children's & Women's Hospital Long Beach, Long Beach, California
  - Velocity Clinical Research - North Hollywood, North Hollywood, California
  - The Neurology Group, Pomona, California
  - UC Davis Medical Center, Investigational Drug Service (IDS) Pharmacy, Sacramento, California
  - University of California, Davis Clinical and Translational Science Center Clinical Research Center, Sacramento, California
  - University of California, Davis Midtown Clinic, Sacramento, California
  - Velocity Clinical Research- Banning, San Bernardino, California
  - Pacific Clinical Research Management Group LLC, Upland, California
  - Sunwise Clinical Research, Walnut Creek, California
  - Children's Hospital Colorado- Investigational Drug Services, Aurora, Colorado
  - Children's Hospital Colorado, Aurora, Colorado
  - Colorado Springs Neurological Associates, PC, Colorado Springs, Colorado
  - Boeson Research GJT, Grand Junction, Colorado
  - Dinosaur Pediatrics, Grand Junction, Colorado
  - CT Clinical Research, Cromwell, Connecticut
  - Ki Health Partners, LLc, dba New England Institute for Clinical Research, Stamford, Connecticut
  - Children's National Medical Center, Washington D.C., District of Columbia
  - AppleMed Research Group, LLC, Miami, Florida
  - Medical Research Center of Miami II, Inc, Miami, Florida
  - South Florida Research Phase I-IV, Inc, Miami Springs, Florida
  - Physicians Group Services, PA d/b/a Coastal Health Research, Orange Park, Florida
  - Clinical Associates of Orlando, LLC, Orlando, Florida
  - ForCare Clinical Research, Tampa, Florida
  - Premiere Research Institute at Palm Beach Neurology, West Palm Beach, Florida
  - Childrens Healthcare of Atlanta, Atlanta, Georgia
  - Rare Disease Research LLC, Atlanta, Georgia
  - Pivotal Clinical Research & Associates, LLC, Brunswick, Georgia
  - CenExel iResearch, LLC, Decatur, Georgia
  - Chicago Headache Center & Research Institute, Chicago, Illinois
  - AMR-Baber Research Inc, Naperville, Illinois
  - Options Research Group, LLC, Westfield, Indiana
  - Integrated Clinical Trial Services, West Des Moines, Iowa
  - Clinical Associates Midwest, LLC, Kansas City, Kansas
  - University of Kentucky Hospital, Lexington, Kentucky
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - MedVadis Research Corporation, Waltham, Massachusetts
  - Michigan Head Pain and Neurological Institute, Ann Arbor, Michigan
  - Corewell Health, for and on behalf of Spectrum Health Hospital and Corewell Health Medical Group, Grand Rapids, Michigan
  - Corewell Health, Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Wellnow Urgent Care and Research, Kalamazoo, Michigan
  - Beaumont Hospital, Royal Oak Campus, Royal Oak, Michigan
  - Sharlin Health Neuroscience Research Center, Ozark, Missouri
  - Clinvest Research, LLC, Springfield, Missouri
  - Boeson Research, Great Falls, Montana
  - Heart & Hands Midwifery, Kalispell, Montana
  - Blue Moose Pediatrics, Missoula, Montana
  - Boeson Research Laboratory, Missoula, Montana
  - Boeson Research, Missoula, Montana
  - Alivation Research, LLC, Lincoln, Nebraska
  - Children's Hospital & Medical Center, Omaha, Nebraska
  - HMH Jersey Shore University Medical Center, Neptune City, New Jersey
  - Dent Neurosciences Research Center, Amherst, New York
  - True North Neurology, Commack, New York
  - New York Neurology Associates, New York, New York
  - Mount Sinai Hospital - Pharmacy Department, New York, New York
  - Columbia University Irving Medical Center, New York, New York
  - Irving Center for Clinical and Translational Research, Outpatient Clinical Research Unit, New York, New York
  - The Neurological Institute of New York, New York, New York
  - North Suffolk Neurology, Port Jefferson Station, New York
  - OnSite Clinical Solutions, LLC, Charlotte, North Carolina
  - Headache Wellness Center, PC, Greensboro, North Carolina
  - WellNow Urgent Care and Research, Cincinnati, Ohio
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - Velocity Clinical Research - Cincinnati, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Wellnow Urgent Care and Research, Dayton, Ohio
  - IPS Research Company, Oklahoma City, Oklahoma
  - Velocity Clinical Research, Grants Pass, Grants Pass, Oregon
  - Providence Brain & Spine Institute-research coordinator's office, Portland, Oregon
  - Providence Health & Services Investigational Drug Services Westside, Portland, Oregon
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Clario, Philadelphia, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Velocity Clinical Research-Providence, East Greenwich, Rhode Island
  - Velocity Clinical Research- Greenville, Greenville, South Carolina
  - Premier Neurology, Greer, South Carolina
  - Novaceut Clinical Research, Clarksville, Tennessee
  - Le Bonheur Children's Hospital, Memphis, Tennessee
  - Le Bonheur Childrens Hospital - Childrens Foundation Research Institute, Memphis, Tennessee
  - Le Bonheur Childrens Hospital - Outpatient Building, Memphis, Tennessee
  - Access Clinical Trials, Inc., Nashville, Tennessee
  - Dell Children's Medical Center, Austin, Texas
  - Child Neurology Consultants of Austin - South Austin, Austin, Texas
  - Child Neurology Consultants of Austin - Central Austin, Austin, Texas
  - Houston Clinical Trials, LLC, Bellaire, Texas
  - Infinite Research Group, LLC, Dallas, Texas
  - Cedar Health Research, Dallas, Texas
  - ANESC Research, El Paso, Texas
  - North Texas Institute of Neurology and Headache, Frisco, Texas
  - Trio Clinical Trials, LLC., Houston, Texas
  - Pain and Headache Centers of Texas, Houston, Texas
  - SCLA Management, Houston, Texas
  - Houston Clinical Research,LLC., Houston, Texas
  - NeuroCare Plus, Houston, Texas
  - AIM Trials, LLC, Plano, Texas
  - JBR Clinical Research, Salt Lake City, Utah
  - Wasatch Clinical Research , LLC(Administrative Location), Salt Lake City, Utah
  - Pediatric Associates of Charlottesville, PLC (Private Pediatric Practice), Charlottesville, Virginia
  - Pediatric Research of Charlottesville, LLC (Regulatory Only), Charlottesville, Virginia
  - Pediatric Research of Charlottesville, LLC, Charlottesville, Virginia
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Children's Specialty Group, PLLC , Division of Childhood & Adolescent Neurology, Norfolk, Virginia
  - National Clinical Research, Inc., Richmond, Virginia
  - Northwest Clinical Research Center, Bellevue, Washington
  - Seattle Children's Hospital Investigational Drug Services, Seattle, Washington
  - Seattle Children's Hospital, Seattle, Washington
  - University Hospital, Madison, Wisconsin
- Poland (6):
  - NZOZ Wielospecjalistyczna Poradnia Lekarska SYNAPSIS, Lech Szczechowski, Katowice
  - Centrum Medyczne Plejady, Krakow
  - Wojewodzki Specjalistyczny Szpital Dzieciecy im. Sw. Ludwika w Krakowie Oddzial Kliniczny Dzieci, Krakow
  - Clinical Research Center Sp. z o.o., Poznan
  - Pracownia Badan Klinicznych SALUS, Wroclaw
  - Centrum Medyczne Oporow, Wroclaw
- Spain (4):
  - Centre Atencio Primaria (CAP) Balenya, Balenya, Barcelona
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Clinico Universitario de Valladolid, Valladolid

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=BHV3000-312